CLINICAL TRIAL: NCT02750579
Title: Early or Delayed Revascularization for Intermediate and High-risk Non ST-elevation Acute Coronary Syndromes?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-A00379-42
Record Dates: First submitted 2016-04-21; First posted 2016-04-25 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): control group: Percutaneous coronary intervention for revascularization delayed intervention (12 to 72 hours)
  Interventions: Procedure: Percutaneous coronary intervention for revascularization
- experimental group (Experimental): experimental group: early Percutaneous coronary intervention for revascularization intervention (<2 hours)
  Interventions: Procedure: Percutaneous coronary intervention for revascularization

INTERVENTIONS:
Procedure: Percutaneous coronary intervention for revascularization — Percutaneous coronary intervention for revascularization with anticoagulant and antiplatelet therapy (routine care)

SUMMARY:
Percutaneous coronary intervention (PCI) is the cornerstone of the care of intermediate and high-risk non ST-elevation acute coronary syndromes (NSTE ACS). Revascularization reduces the rate of cardiovascular death and recurrent myocardial infarction in this clinical setting. The recommendation regarding the timing of intervention in this clinical setting is derived from old trials and has a weak level of evidence. In fact, there are no conclusive randomized trials in the contemporary era providing guidance on the optimal timing of intervention. In addition, the optimal timing of this critical intervention has not been studied since the development of new P2Y12-ADP receptor antagonists and the controversy surrounding the use of pretreatment with a P2Y12-ADP receptor antagonist before intervention. Early intervention in intermediate and high-risk non ST-elevation ACS is not well validated to date. In addition, the recent changes in the use of pretreatment with P2Y12-ADP receptor antagonists may impact on the potential benefit of an early intervention.

Based on these evidences, we hypothesize that with the current protocols of care without pretreatment with a P2Y12-ADP receptor antagonist, an early PCI (<2 hours) would be superior to a delayed (between 12 to 72 hours) PCI in the setting of intermediate or high-risk non-ST elevation acute coronary syndrome to prevent cardiovascular death and ischemic recurrences.

ELIGIBILITY:
Inclusion Criteria:

* Must not be of child-bearing potential (1 year post-menopausal, contraceptive use or surgically sterile);
* Subject with a non-ST-segment elevation ACS defined by the presence of at least 2 of the following criteria: symptoms of myocardial ischemia, electrocardiographic ST-segment abnormalities (depression or transient elevation of at least 0.1 mV) or T-wave inversion in at least in 2 contiguous leads, or an elevated cardiac troponin value (above the upper limit of normal) ;
* Subject requiring intervention according to physician's judgment including the following criteria subject with one of the following risk factor defining intermediate and high risk ACS: diabetes mellitus, kidney failure, reduced LVEF, early post infarction angina, recent PCI, prior CABG or a GRACE risk score >109, recurrent symptoms or ischaemia on non-invasive testing (2);
* Must be enrolled at a cardiac catheterization laboratory hospital or at a hospital/ambulance service affiliated with a cardiac catheterization laboratory hospital;

Exclusion Criteria:

* - Minors or pregnant or breast-feeding women;
* Subject with low risk ACS;
* Subject with very high-risk ACS: refractory angina, severe heart failure, life-threatening ventricular arrhythmias, hemodynamic instability requiring immediate intervention;
* Subject with thrombolytic therapy during the preceding 24 hours;
* Subject with bleeding diathesis;
* Subject with Upstream treatment by a GPIIb/IIIa inhibitor;
* Subject under chronic anticoagulant;
* Subject participating in another research protocol;
* Subject not agreeing to participate;
* Subject with contraindication to or under chronic P2Y12 receptor antagonists therapy (clopidogrel, ticagrelor and prasugrel);
* Present with ST-segment elevation myocardial infarction (STEMI) at the time of entry or randomization into the study defined as follows:
* ST-segment elevation myocardial infarction is defined as a history of chest discomfort or ischemic symptoms of >20 minutes duration at rest ≤14 days prior to entry into the study with one of the following present on at least one ECG prior to randomization:

  1. ST-segment elevation ≥1 mm in two or more contiguous ECG leads.
  2. New or presumably new left bundle branch block (LBBB).
  3. ST-segment depression ≥1 mm in two anterior precordial leads (V1 through V4) with clinical history and evidence suggestive of true posterior infarction.
* Have cardiogenic shock (systolic blood pressure <90 mm Hg associated with clinical evidence of end-organ hypoperfusion, or subjects requiring vasopressors to maintain systolic blood pressure over 90 mm Hg and associated with clinical evidence of end-organ hypoperfusion);
* Have New York Heart Association (NYHA) Class IV congestive heart failure (CHF).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 740 (Actual)
Dates: Start 2016-09-05 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
recurrent ischemic events | 1 month
  compare the efficacy defined by the rate of recurrent ischemic events at 1 month of 2 therapeutic strategies: an immediate (<2 hours) versus a delayed (12-72 hours) intervention for intermediate and high-risk non ST-elevation acute coronary syndrome compare the efficacy defined by the rate of cardiovascular death and/or recurrent ischemic events at 1 month of 2 therapeutic strategies: an immediate (<2 hours) versus a delayed (12-72 hours) intervention for intermediate and high-risk non ST-elevation acute coronary syndrome
cardiovascular death | 1 month
  compare the efficacy defined by the rate of cardiovascular death at 1 month of 2 therapeutic strategies: an immediate (<2 hours) versus a delayed (12-72 hours) intervention for intermediate and high-risk non ST-elevation acute coronary syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Bonello, MD, Principal Investigator — assistance Public Hopitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lemesle G, Laine M, Pankert M, Boueri Z, Motreff P, Paganelli F, Baumstarck K, Roch A, Kerbaul F, Puymirat E, Bonello L. Optimal Timing of Intervention in NSTE-ACS Without Pre-Treatment: The EARLY Randomized Trial. JACC Cardiovasc Interv. 2020 Apr 27;13(8):907-917. doi: 10.1016/j.jcin.2020.01.231. PMID 32327087
- [Derived] Lemesle G, Laine M, Pankert M, Puymirat E, Bonello L. Great expectations. Lancet. 2018 Jan 27;391(10118):306. doi: 10.1016/S0140-6736(18)30096-5. Epub 2018 Jan 31. No abstract available. PMID 29413039